CLINICAL TRIAL: NCT06844955
Title: Impact of Using a Smart Diabetic Foot Care Application on Patients' Knowledge and Self-management
Brief Title: Smart Diabetic Foot Care Application
Acronym: NTUNHS
Status: Active, not recruiting | Type: Observational
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Pei-Hung Liao, Professor, National Taipei University of Nursing and Health Sciences
Other Study IDs: 112-058B
Record Dates: First submitted 2025-02-11; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Vital signs measurement data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study developed an app for the guidance of home-based diabetic foot care to explore its impact on patients' foot assessment awareness and self-care behavior after using this app. The study also assessed the app's effectiveness in cultivating behavioral habits that are effective in managing diabetes.

DETAILED DESCRIPTION:
Diabetes is a common chronic metabolic disease worldwide. Approximately 50% to 60% of ulcers caused by diabetes become infected, and moderate to severe infections can lead to lower limb amputation. Among amputees, the five-year mortality rate exceeds 70%.Smart devices (mobile phones, computers, etc.) are indispensable necessities to modern lives. Downloadable mobile health applications (mHealth Apps) on smartphones are widely used in medical care . The use of these apps on smartphones has created a new field in the health industry known as mobile health

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 2 diabetes .
2. Aged between 20 and 80 years.
3. Able to use mobile apps or tablets for health management .

Exclusion Criteria:

1. Patients who were unconscious, had delirium, were bedridden, had cognitive impairment, or were unable to perform daily self-care.
2. Patients who refused to participate.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Collect diabetes cases from a Christian hospital in the northeast that agrees to join this program
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Foot ulcers | 3 months
  This study collest Vital signs data and used questionnaires to collect data on whether patients had certain types of chronic diseases, whether they exercised regularly, and on medication use. In addition to diabetes, other chronic conditions, including hypertension, respiratory diseases, heart disease, urinary system disorders, immune system diseases, and hyperlipidemia, were also considered. The study took chronic diseases, exercise, and medication as independent variables. Logistic regression analysis of the association and risk estimation for foot ulcers

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei university of nursing and health science, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided